CLINICAL TRIAL: NCT05925023
Title: Sirolimus in the Treatment of Refractory/Relapsed Warm Autoimmune Hemolytic Anemia (AIHA)： a Phase 2 Prospective Trial
Brief Title: Sirolimus in the Treatment of Refractory/Relapsed wAIHA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Chen Miao, associate professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sirolimus-1
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Warm Autoimmune Hemolytic Anemia
Keywords: warm autoimmune hemolytic anemia; Evans syndrome; refractory/relapsed; sirolimus; efficacy
MeSH Terms: conditions — Evans Syndrome; Recurrence | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sirolimus on refractory/relapsed wAIHA (Experimental): A prospective research of the sirolimus efficiency on refractory/relapsed primary wAIHA patients. Sirolimus dosage: 1-3 mg/d with plasma concentration 4-15ng/mL. Medication time should last at least 6 months. After reaching the optimal response, responders continue to use sirolimus for 1 year, and then gradually reduce the dosage.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Oral administration, 1-3 mg/d, sirolimus plasma concentration: 4-15 ng/mL

SUMMARY:
Autoimmune hemolytic anemia (AIHA) is a rare and heterogeneous disorder characterized by the destruction of red blood cells through warm or cold antibodies. Glucocorticoid (combined with rituximab) is the first-line treatment. However, the recurrence rate is very high and some patients may not respond to steroids. Second-line therapies include cyclosporine A (CsA), cyclophosphamide, rituximab, azathioprine, and even splenectomy. Our previous study of sirolimus in refractory/relapsed AIHA and ES found an effective rate of 80%. Therefore, the investigators plan to explore the efficacy and safety of sirolimus in the treatment of refractory/relapsed wAIHA.

DETAILED DESCRIPTION:
Based on the optimal autoantibody-RBC reactivity temperatures, AIHA is classified into warm type, cold type, and mixed type. AIHA can be further classified into primary or secondary in nature. Glucocorticoid (combined with rituximab) is the first-line treatment. However, the recurrence rate is very high and some patients may not respond to steroids. Second-line therapies include cyclosporine A (CsA), cyclophosphamide, rituximab, azathioprine, and even splenectomy. The refractory/relapsed wAIHA patients have increased cardiovascular events, increased opportunities for infections, decreased quality of life, and even death. A prospective multi-institutional trial in autoimmune cytopenia found that 8 of 10 patients with AIHA and Evans syndrome respond to sirolimus. Our previous study of sirolimus in refractory/relapsed AIHA and ES also found an effective rate of approximately 80%. Since sirolimus is cheap and accessible, our findings may reduce the economic burden of patients and be a guide on the selection of second-line treatment drugs in refractory/relapsed wAIHA and Evans syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. Diagnosed as primary warm autoimmune hemolytic anemia or Evans syndrome (primary or secondary). There is no treatment indication of other systemic involvement in the original disease if secondary.
3. No response to glucocorticoid therapy or recurrence.
4. Baseline liver (ALT, AST) was less than 2 times the normal value.
5. No active infection; Not pregnant or breastfeeding.
6. Agree to sign the consent form.

Exclusion Criteria:

1. Patients with connective tissue disease or other organs involvement
2. Infection or bleeding that cannot be controlled by standard treatment.
3. Active HIV, HCV or HBV infection or cirrhosis or portal hypertension.
4. Progressed uncontrolled malignant tumors and lymphoma
5. Cirrhosis or portal hypertension.
6. Pregnant or breastfeeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-06-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) and complete response rate (CRR) | 3,6,12 months
  ORR defined as the proportion of patients who met the criteria of either complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events and the number of relapses | 12 months, end of the follow-up
  Number of participants with treatment-related adverse events and the number of relapses
Adverse events | 3,6,12 months
  Safety analyses include assessments of the incidence and severity of adverse events; all adverse events that occurred or worsened during the treatment period will be reported, as well as adverse events that occurred later but are considered by the investigator to be related to the trial drug.
Relapse rate | 3,6,12 months
  Relapse rate defined as the proportion of patients whose response shift from PR or CR to no response (NR).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jager U, Barcellini W, Broome CM, Gertz MA, Hill A, Hill QA, Jilma B, Kuter DJ, Michel M, Montillo M, Roth A, Zeerleder SS, Berentsen S. Diagnosis and treatment of autoimmune hemolytic anemia in adults: Recommendations from the First International Consensus Meeting. Blood Rev. 2020 May;41:100648. doi: 10.1016/j.blre.2019.100648. Epub 2019 Dec 5. PMID 31839434
- [Background] Bass GF, Tuscano ET, Tuscano JM. Diagnosis and classification of autoimmune hemolytic anemia. Autoimmun Rev. 2014 Apr-May;13(4-5):560-4. doi: 10.1016/j.autrev.2013.11.010. Epub 2014 Jan 11. PMID 24418298
- [Background] Hill QA, Stamps R, Massey E, Grainger JD, Provan D, Hill A; British Society for Haematology. The diagnosis and management of primary autoimmune haemolytic anaemia. Br J Haematol. 2017 Feb;176(3):395-411. doi: 10.1111/bjh.14478. Epub 2016 Dec 22. No abstract available. PMID 28005293
- [Background] Barcellini W, Fattizzo B. How I treat warm autoimmune hemolytic anemia. Blood. 2021 Mar 11;137(10):1283-1294. doi: 10.1182/blood.2019003808. PMID 33512406
- [Background] Birgens H, Frederiksen H, Hasselbalch HC, Rasmussen IH, Nielsen OJ, Kjeldsen L, Larsen H, Mourits-Andersen T, Plesner T, Ronnov-Jessen D, Vestergaard H, Klausen TW, Schollkopf C. A phase III randomized trial comparing glucocorticoid monotherapy versus glucocorticoid and rituximab in patients with autoimmune haemolytic anaemia. Br J Haematol. 2013 Nov;163(3):393-9. doi: 10.1111/bjh.12541. Epub 2013 Aug 24. PMID 23981017
- [Background] Barcellini W, Fattizzo B, Zaninoni A, Radice T, Nichele I, Di Bona E, Lunghi M, Tassinari C, Alfinito F, Ferrari A, Leporace AP, Niscola P, Carpenedo M, Boschetti C, Revelli N, Villa MA, Consonni D, Scaramucci L, De Fabritiis P, Tagariello G, Gaidano G, Rodeghiero F, Cortelezzi A, Zanella A. Clinical heterogeneity and predictors of outcome in primary autoimmune hemolytic anemia: a GIMEMA study of 308 patients. Blood. 2014 Nov 6;124(19):2930-6. doi: 10.1182/blood-2014-06-583021. Epub 2014 Sep 16. PMID 25232059
- [Background] Bride KL, Vincent T, Smith-Whitley K, Lambert MP, Bleesing JJ, Seif AE, Manno CS, Casper J, Grupp SA, Teachey DT. Sirolimus is effective in relapsed/refractory autoimmune cytopenias: results of a prospective multi-institutional trial. Blood. 2016 Jan 7;127(1):17-28. doi: 10.1182/blood-2015-07-657981. Epub 2015 Oct 26. PMID 26504182
- [Background] Li H, Ji J, Du Y, Huang Y, Gu H, Chen M, Wu R, Han B. Sirolimus is effective for primary relapsed/refractory autoimmune cytopenia: a multicenter study. Exp Hematol. 2020 Sep;89:87-95. doi: 10.1016/j.exphem.2020.08.001. Epub 2020 Aug 6. PMID 32771553